CLINICAL TRIAL: NCT06773273
Title: A Novel Approach to Lens Subluxation: CapsuLaser and Flanged Prolene Suture for Cionni Ring Scleral Fixation
Brief Title: A Novel Approach to Lens Subluxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEH-IRB# 355 -5-January -2025; Maghrabi eye hospitals (Other: Zagazig university)
Record Dates: First submitted 2024-12-29; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Subluxation
Keywords: Subluxation, CapsuLaser, Prolene, Cionni
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Intervention Model Description: This retrospective interventional randomized study included 15 eyes of 15 patients; six of them were due to pseudo exfoliation, five of them were males while the other nine cases were due to hereditary lens subluxation eight of them were females.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CapsuLaser-Assisted Capsulorhexis and Flanged Prolene Suture (Other): CapsuLaser-Assisted Capsulorhexis and Flanged 6-0 Prolene Suture for Cionni Ring Scleral Fixation
  Interventions: Procedure: CapsuLaser-Assisted Capsulorhexis and Flanged Prolene Suture

INTERVENTIONS:
Procedure: CapsuLaser-Assisted Capsulorhexis and Flanged Prolene Suture — CapsuLaser-Assisted Capsulorhexis and Flanged 6-0 Prolene Suture for Cionni Ring Scleral Fixation

SUMMARY:
Evaluating new technique for treating patients with subluxation using specific laser type and new 6-0 proline fixating novel technique for the capsular bag

DETAILED DESCRIPTION:
The management of a subluxated crystalline lens remains a challenge for anterior segment surgeons, largely due to the complex anatomical and functional changes in such cases. Capsulaser is safe and effective tool in creating well centered CCC with consistent 360 degree IOL coverage that ensures better lens stability and effective lens positioning . Combined with using flanged 6-0 Prolene sutures for scleral fixation of Cionni rings, this technique addresses previous limitations by improving intraoperative control.

ELIGIBILITY:
Inclusion Criteria:

* Lens subluxation with clear corneal media.

Exclusion Criteria:

* Associated macular lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Number of cases with IOL centration inside the capsular bag | 6 months
  the long term stability of the capsular bag

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMIR, MD,PhD, Principal Investigator — Zagazig University
Locations (1):
- Maghrabi Eye Hospitals, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No